CLINICAL TRIAL: NCT03748849
Title: Is the Subjective Experience of Recovery From Low Back Pain Related a Decrease in the Sensitivity of Pain Mechanisms?
Brief Title: Pain Sensory Profile Changes Following Treatment of Chronic Low Back Pain
Acronym: LBP
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Thorvaldur Skuli Palsson, Assistant professor, Aalborg University
Other Study IDs: N-20150048
Record Dates: First submitted 2018-11-12; First posted 2018-11-21 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain group: Males and females who have had low back pain lasting between 12 weeks - 5 years without any other health problems (physical or psychological). Following baseline measurements, all subjects are offered individualized physiotherapy. The interventions mainly consist of exercises targeting their functional limitations. These are supplemented by a thorough explanation of their pain condition. This is done within the boundaries of the current understanding of musculoskeletal pain. This is supplemented with encouragement to do regular exercise and with manual therapy if needed/indicated.
  Interventions: Procedure: Physiotherapy
- Control group: Healthy males and females who have no current musculoskeletal pain problem (specific to the low back and/or in general). Likewise, they cannot have a previous history of on-going musculoskeletal pain. On-going pain is defined as a condition that limited their function for 3 months or more.
  Participants in the control group take part in the baseline measurement and then another measurement after 6-8 weeks

INTERVENTIONS:
Procedure: Physiotherapy
  Groups: Low back pain group

SUMMARY:
Several cross-sectional studies have demonstrated that patients with chronic low back pain have higher levels of pain sensitivity (local and widespread) when compared to controls. It is unclear however, if improvements in pain and function are reflected in a decrease in the sensitivity of pain mechanisms. This study compares the pain sensory profile in patients with chronic low back pain before and after a period of physiotherapy treatment. To account for natural fluctuations in pain sensitivity, healthy age matched controls are also measured twice

DETAILED DESCRIPTION:
The sensitivity of pain mechanisms has consistently been shown to be increased in people suffering from chronic low back pain. This includes both sensitivity in the painful region but also in areas distant indicating widespread pain sensitivity. It is less clear whether this is normalized following a successful treatment intervention.

This study is recruiting people with low back pain and healthy, age matched controls. At baseline, the following measurements are made:

* the sensitivity to pressure (at the low back and at the shoulder)
* the pain detection threshold and pain tolerance threshold at the lower legs
* the temporal summation of pain
* conditioned pain modulation
* Fear-avoidance beliefs
* Disability (Roland-Morris Disability Questionnaire)
* The Orebro musculoskeletal pain questionnaire

During their enrollment, the patients report their weekly pain electronically

All quantitative sensory testing (QST) and questionnaire data are blind to the principal investigator until data collection has been finished

After the baseline measurements, the patients are offered physiotherapy treatment. The treatment protocol (dosage and type of intervention) is designed based on individual needs following an assessment by a musculoskeletal physiotherapist. The number of sessions and time between treatment sessions depend on how the patients respond to the chosen intervention. Patients are discharged from treatment when:

1. they have made sufficient recovery (their back pain is no longer a problem)
2. the chosen intervention(s) have failed to affect their condition
3. no more recovery is expected

The quantitative sensory testing measurements are performed again after discharge

ELIGIBILITY:
Inclusion Criteria:

Patient group

* Pain located in the low back region, defined as the area lying between the posterior superior iliac spine below and the thoracolumbar junction above
* The pain has lasted between 3 and 60 months

Exclusion Criteria:

* Pain related to a specific pathology such as spinal stenosis, metastasis, fracture etc.
* Leg pain related to nerve root compression/irritation.
* Multiple painful sites/areas unrelated to the back pain
* Operation to the spine
* Any neurological or systemic diseases which can affect the outcome measures
* Pregnancy
* Lack of ability to cooperate

Control group Inclusion Criteria

• Are healthy and free from any pain specific to the low back and/or in general

Exclusion Criteria

* No current or previous history of on-going pain, defined as pain lasting more than 3 months, in the lumbopelvic region and/or elsewhere
* Have participated in studies using a similar experimental pain model

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Low back pain group Males and females who have had low back pain lasting 3 - 60 months. The reason for onset (traumatic/non-traumatic) is registered but not used for inclusion/exclusion
  Control group Healthy males and females with no current or previous history of musculoskeletal pain. Previous history is defined as pain of on-going nature (lasting 3 months or more) in the low back and/or in general
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Change in cuff-pressure mechanical sensitivity, measured with a computer-controlled pressure cuff | At baseline and after discharge from treatment (patients) or after 6-8 weeks (controls)
  The pressure needed to evoke first onset of pain (pain detection threshold, PDT) and the most pressure tolerable (pain tolerance threshold, PTT) are measured with a computer controlled pressure cuff. The cuff is placed on the lower leg and is gradually inflated (1kPa/sec). The first onset of pain (VAS 1, measured on an electronic VAS scale: 0=no pain, 10=worst pain imaginable) is indicated when the sensation of pressure around the leg changes to pain. The pressure continues to rise until the PTT is reached. PTT is defined as the point where the subject cannot endure more increase in pressure.
Sensitivity to mechanical point pressure measured with a handheld pressure algometer | At baseline and after discharge from treatment (patients) or after 6-8 weeks (controls)
  Change in sensitivity to mechanical point pressure back (L5 and L1) and shoulder (infraspinatus) between baseline and discharge from rehabilitation.
  Mechanical point pressure is measured with a handheld pressure algometer (Somedic, Sweden). The average from dominant and non-dominant sides will be used for analysis
Temporal summation of pain (increase in pain from repeated nociceptive stimuli at the same intensity) measured with a computer-controlled pressure cuff | At baseline and after discharge from treatment (patients) or after 6-8 weeks (controls)
  Change in temporal summation of pain between baseline and follow-up. Temporal summation of pain is assessed by using a computer controlled pressure cuff which is mounted on the lower leg on the dominant side. The participant receives 10 stimuli with a 1sec break between stimuli. Immediately following each stimuli, the participants rates the pain intensity using an electronic VAS scale (0-10, where 0=no pain and 10=worst pain imaginable)
Conditioned pain modulation (change in pain sensitivity following the onset of a competing, nociceptive stimulus) measured with a computer-controlled pressure cuff | At baseline and after discharge from treatment (patients) or after 6-8 weeks (controls)
  Change in conditioned pain modulation between baseline and follow-up. Conditioned pain modulation is assessed by using two computer controlled pressure cuffs which are mounted on the lower legs, one on each side. On the non-dominant side, the cuff is inflated rapidly up to 80% of the pain tolerance threshold and kept there steady. In the meanwhile, the pain detection threshold and pain tolerance thresholds are assessed on the dominant side. Changes in PDT and PTT compared with baseline are defined as a CPM response.

SECONDARY OUTCOMES:
Pain (measured on a numeric rating scale) | At baseline and after discharge from treatment (patients) or after 6-8 weeks (controls)
  Change in pain between baseline and follow-up measured on a numeric rating scale (0 = no pain and 10 = worst pain imaginable)
Disability measured on the Roland-Morris Disability Questionnaire | At baseline and after discharge from treatment (patients) or after 6-8 weeks (controls)
  Change in disability between baseline and follow-up will be found by comparing baseline measurements with measurements at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health Science and Technology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No